CLINICAL TRIAL: NCT03697109
Title: Glucocorticoid Receptor Antagonism in the Treatment of Cushing Syndrome (GRACE): A Phase 3, Double-Blind, Placebo-Controlled, Randomized-Withdrawal Study of the Efficacy and Safety of Relacorilant
Brief Title: A Study of the Efficacy and Safety of Relacorilant in Patients With Endogenous Cushing Syndrome
Acronym: GRACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CORT125134-455
Record Dates: First submitted 2018-09-27; First posted 2018-10-05 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-04

CONDITIONS: Cushing Syndrome
Keywords: Cushing syndrome; Cushing disease; Hypercortisolemia; Cushingoid; Type 2 Diabetes; Impaired Glucose Intolerance; Hypertension; Adrenocorticotropic hormone; Primary Pigmented Nodular Adrenal Disease; Moon Facies; Dorsocervical Fat Pad; Adrenal Adenoma; Adrenal Autonomy; Cortisol; Cushing
MeSH Terms: conditions — Cushing Syndrome; Pituitary ACTH Hypersecretion; ACTH Syndrome, Ectopic; Diabetes Mellitus, Type 2; Hypertension | interventions — relacorilant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Relacorilant (OL Phase) (Experimental): Patients will receive relacorilant increased sequentially from 100 mg once daily to a maximum dose of 400 mg once daily.
  Interventions: Drug: Relacorilant
- Relacorilant (RW Phase) (Experimental): Patients who meet any of the response criteria will advance to the RW Phase of the study and receive the same dose of relacorilant as the last dose administered in the OL Phase.
  Interventions: Drug: Relacorilant
- Placebo (RW Phase) (Placebo Comparator): Patients who meet any of the response criteria will advance to the RW Phase of the study and receive placebo matched to study drug.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Relacorilant — Relacorilant is supplied as 100 mg capsules for oral dosing.
  Other Names: CORT125134
  Arms: Relacorilant (OL Phase); Relacorilant (RW Phase)
Other: Placebo — Placebo matched to study drug
  Arms: Placebo (RW Phase)

SUMMARY:
This is a Phase 3, double-blind, placebo-controlled, randomized-withdrawal study to assess the efficacy, safety and pharmacokinetics (PK) of relacorilant in patients with endogenous Cushing syndrome and concurrent type 2 diabetes mellitus/impaired glucose tolerance (DM/IGT) and/or uncontrolled hypertension (HTN).

DETAILED DESCRIPTION:
The primary outcome is the assessment of efficacy of relacorilant treatment based on sustained blood pressure control during the Randomized-withdrawal (RW) Phase, wherein patients who had achieved the blood pressure response criteria during the Open-label (OL) Phase are randomized to receive either relacorilant or placebo for 12 weeks.

Patients in the OL Phase will dose-escalate in 100 mg increments to a maximum dose of 400 mg orally once daily. Patients will remain on OL treatment until Week 22 at which time they will be evaluated for the RW Phase based on predefined hyperglycemia and hypertension response criteria. Eligible patients will then be randomized to receive either relacorilant or placebo at a 1:1 ratio for 12 weeks. Patients who do not meet the criteria for the RW Phase will end treatment and may be eligible to roll over into an extension safety study. Patients who complete the RW Phase of the study may also be eligible to roll over into an extension study.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed diagnosis of endogenous Cushing syndrome
* Meets at least 1 of the following criteria:

  * Has Type 2 diabetes mellitus
  * Has impaired glucose tolerance
  * Has hypertension.

Exclusion Criteria:

* Has non-endogenous source of hypercortisolism
* Has uncontrolled, clinically significant hypothyroidism or hyperthyroidism
* Has poorly controlled hypertension
* Has poorly controlled diabetes mellitus
* Has severe renal insufficiency.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Moraitis, MD, Study Director — Corcept Therapeutics
Locations (64):
- United States (32):
  - Site 21, Phoenix, Arizona
  - Site 36, Los Angeles, California
  - Site 68, Torrance, California
  - Site 10, Miami, Florida
  - Site 14, Atlanta, Georgia
  - Site 41, Chicago, Illinois
  - Site 7, Indianapolis, Indiana
  - Site 2, Metairie, Louisiana
  - Site 45, Baltimore, Maryland
  - Site 46, Boston, Massachusetts
  - Site 20, Ann Arbor, Michigan
  - Site 4, Jackson, Mississippi
  - Site 13, St Louis, Missouri
  - Site 53, Omaha, Nebraska
  - Site 72, Reno, Nevada
  - Site 8, Albany, New York
  - Site 6, Jamaica, New York
  - Site 57, New York, New York
  - Site 35, New York, New York
  - Site 39, New York, New York
  - Site 1, Wilmington, North Carolina
  - Site 17, Columbus, Ohio
  - Site 11, Oklahoma City, Oklahoma
  - Site 62, Philadelphia, Pennsylvania
  - Site 19, Pittsburgh, Pennsylvania
  - Site 71, Pittsburgh, Pennsylvania
  - Site 5, Summerville, South Carolina
  - Site 51, Dallas, Texas
  - Site 3, El Paso, Texas
  - Site 65, Houston, Texas
  - Site 56, Shavano Park, Texas
  - Site 31, Everett, Washington
- Site 47, Vienna, Austria
- Site 27, Sofia, Bulgaria
- Canada (2):
  - Site 70, Halifax, Nova Scotia
  - Site 58, Montreal
- Germany (2):
  - Site 54, München
  - Site 49, Würzburg
- Israel (4):
  - Site 30, Jerusalem
  - Site 29, Kfar Saba
  - Site 28, Petah Tikva
  - Site 69, Tel Aviv
- Italy (8):
  - Site 43, Ancona
  - Site 15, Messina
  - Site 26, Milan
  - Site 12, Napoli
  - Site 38, Orbassano
  - Site 67, Padua
  - Site 40, Roma
  - Site 16, Roma
- Site 34, Rotterdam, Netherlands
- Poland (4):
  - Site 77, Bialystok
  - Site 37, Chrzanów
  - Site 59, Krakow
  - Site 33, Lublin
- Romania (4):
  - Site 66, Bucharest
  - Site 63, Bucharest
  - Site 64, Bucharest
  - Site 73, Iași
- Spain (5):
  - Site 75, Alicante
  - Site 25, Girona
  - Site 24, Madrid
  - Site 22, Málaga
  - Site 23, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pivonello R, Munster PN, Terzolo M, Ferrigno R, Simeoli C, Puglisi S, Bali U, Moraitis AG. Glucocorticoid Receptor Antagonism Upregulates Somatostatin Receptor Subtype 2 Expression in ACTH-Producing Neuroendocrine Tumors: New Insight Based on the Selective Glucocorticoid Receptor Modulator Relacorilant. Front Endocrinol (Lausanne). 2022 Jan 4;12:793262. doi: 10.3389/fendo.2021.793262. eCollection 2021. PMID 35058882

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 404 patients were screened and 152 were enrolled.
Period: Open-label (OL) Phase
Arm/Group | Relacorilant (OL Phase) | Relacorilant (RW Phase) | Placebo (RW Phase)
Started | 152 | 0 | 0
Completed | 95 | 0 | 0
Not Completed | 57 | 0 | 0
Not completed — Adverse Event | 24 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Lack of Efficacy | 6 | 0 | 0
Not completed — Withdrawal by Subject | 21 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Death | 2 | 0 | 0
Period: Randomized-withdrawal (RW) Phase
Arm/Group | Relacorilant (OL Phase) | Relacorilant (RW Phase) | Placebo (RW Phase)
Started | 0 | 30 | 32
Completed | 0 | 27 | 31
Not Completed | 0 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The analysis population was patients in the Intent-to-Treat (ITT) Population which included all enrolled patients who received at least 1 dose of study drug.
Arm/Group | Relacorilant (OL Phase)
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 123
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 18
  White | 121
  More than one race | 6
  Unknown or Not Reported | 6
Body weight [Mean (Standard Deviation); unit: kg] | 93.77 (24.660)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.738 (32.675)
Waist circumference [Mean (Standard Deviation); unit: cm] | 114.85 (18.0355)
Hypertension (HTN) only [Count of Participants; unit: Participants] — HTN is defined as mean systolic blood pressure (SBP) ≥135 or ≤170 mm Hg and/or mean diastolic blood pressure (DBP) ≥85 to ≤110 mm Hg.
  Participants | 31
Diabetes mellitus (DM) or impaired glucose tolerance (IGT) only [Count of Participants; unit: Participants] — DM is defined as fasting plasma glucose ≥126 mg/dL and/or oral glucose tolerance test plasma glucose ≥200 mg/dL or hemoglobin A1c (HbA1c) ≥6.5%. IGT is defined as plasma glucose ≥140 mg/dL and <200 mg/dL on a 2-hour oral glucose tolerance test.
  Participants | 50
HTN and DM/IGT [Count of Participants; unit: Participants] — HTN and DM/IGT as previously defined.
  Participants | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Loss of Response With Respect to Hypertension During the RW Phase.
Description: Loss of response with respect to HTN was measured using 6 criteria: 1) an increase in SBP of at least 5 mm Hg, 2) an increase in DBP of at least 5 mm Hg, 3) an increase in SBP and/or DBP of at least 5 mm Hg, 4) use of HTN rescue medication, 5) treatment discontinuation, and 6) missing 24-hour ambulatory blood pressure monitoring (ABPM) measurement at the end of the RW Phase. Blood pressure was measured using ABPM. Use of rescue medication was defined as any increase, modification, or addition of antihypertensive medication due to worsening HTN. Treatment discontinuation reports the number of patients who discontinued study treatment in the RW Phase for any reason.
Time Frame: Week 22 (end of OL Phase) and Week 36 (Week 12 of RW Phase)
Population: The analysis population was patients in the Intent-to-Treat (ITT-RW) Population who met the HTN response criteria at conclusion of the OL Phase. The ITT-RW Population included all patients who were randomized in the RW Phase and received at least 1 dose of study drug post randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant (RW Phase) | Placebo (RW Phase)
Number analyzed (Participants) | 21 | 22
Participants
  SBP | 3 | 1
  DBP | 1 | 1
  SBP and/or DBP | 3 | 4
  Use of rescue medication | 0 | 7
  Treatment discontinuation | 2 | 3
  Missing ABPM at end of RW Phase | 2 | 3
Statistical Analysis 1: Comparison: Relacorilant (RW Phase) vs Placebo (RW Phase); A logistic regression model with logit link function was used in order to detect if there was a significant difference in total number of patients with a loss of response with respect to HTN under treatment with relacorilant compared with treatment with placebo in the RW Phase; Test type: Equivalence — Log odds is equal to 0 (null hypothesis) vs log odds not equal to 0 (alternative hypothesis); p = 0.0215, Chi-squared; Odds Ratio (OR) = 0.17, 95% CI 2-sided [0.04 to 0.77] — An odds ratio (OR) <1 represents lower odds of loss of response under treatment with relacorilant compared with treatment with placebo

2. Primary Outcome: Number of Patients With 1 or More Treatment-emergent Adverse Events (TEAEs) as Graded by CTCAE v5.0.
Time Frame: OL Phase: Up to 22 weeks; RW Phase: up to 18 weeks after completion of the OL Phase
Population: The analysis population was patients in the Safety Population, which included all enrolled patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant (OL Phase) | Relacorilant (RW Phase) | Placebo (RW Phase)
Number analyzed (Participants) | 152 | 30 | 32
Participants | 147 | 23 | 27

3. Secondary Outcome: Change in Area Under the Concentration-time Curve of Blood Glucose (AUCglucose) During the RW Phase
Time Frame: Before and at time intervals up to 2 hours post glucose drink at Week 22 (end of OL Phase) and Week 36 (Week 12 of RW Phase)
Population: The analysis population was patients in the ITT-RW Population who had DM/IGT with or without HTN at Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: hours x mmol/L
Arm/Group | Relacorilant (RW Phase) | Placebo (RW Phase)
Number analyzed (Participants) | 18 | 20
hours x mmol/L | 1.91 [-1.138 to 4.966] | 4.81 [2.096 to 7.529]

4. Secondary Outcome: Change in Hemoglobin HbA1c During the RW Phase
Time Frame: Week 22 (end of OL Phase) and Week 36 (Week 12 of RW Phase)
Population: The analysis population was patients in the ITT-RW Population who had DM/IGT with or without HTN at Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Relacorilant (RW Phase) | Placebo (RW Phase)
Number analyzed (Participants) | 16 | 19
Percentage | 0.06 [-0.270 to 0.383] | 0.28 [-0.022 to 0.578]

5. Secondary Outcome: Change in 2-hour Plasma Glucose During the RW Phase
Description: Plasma glucose was measured using the 2-hour Oral Glucose Tolerance Test (oGTT).
Time Frame: Before and 2 hours post glucose drink at Week 22 (end of OL Phase) and Week 36 (Week 12 of RW Phase)
Population: The analysis population was patients in the ITT-RW Population who had DM/IGT with or without HTN at Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Relacorilant (RW Phase) | Placebo (RW Phase)
Number analyzed (Participants) | 15 | 19
mmol/L | 0.52 [-1.06 to 2.09] | 2.96 [1.55 to 4.37]

6. Secondary Outcome: Change in SBP and DBP During the RW Phase
Description: Blood pressure was measured by 24-hour ABPM.
Time Frame: Week 22 (end of OL Phase) and Week 36 (Week 12 of RW Phase)
Population: The analysis population was patients in the ITT-RW Population who had HTN with or without DM/IGT at Baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Relacorilant (RW Phase) | Placebo (RW Phase)
Number analyzed (Participants) | 21 | 22
mm Hg
  SBP | 3.95 [0.470 to 7.424] | 10.43 [6.538 to 14.329]
  DBP | 2.86 [-0.199 to 5.928] | 6.53 [3.224 to 9.832]

7. Secondary Outcome: Change in Body Weight During the RW Phase
Time Frame: Week 22 (end of OL Phase) and Week 36 (Week 12 of RW Phase)
Population: The analysis population was patients in the ITT-RW Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Relacorilant (RW Phase) | Placebo (RW Phase)
Number analyzed (Participants) | 26 | 30
kg | -1.21 [-2.685 to 0.269] | 0.54 [-0.851 to 1.939]

8. Secondary Outcome: Number of Patients With Any Increase or Modification in Diabetes Medication During the RW Phase
Time Frame: Week 22 (end of OL Phase) and up to Week 36 (Week 12 of RW Phase)
Population: The analysis population was patients in the ITT-RW Population who had DM/IGT at Baseline and received antidiabetic medication during the RW Phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Relacorilant (RW Phase) | Placebo (RW Phase)
Number analyzed (Participants) | 7 | 8
Participants | 1 | 0

9. Other Pre Specified Outcome: Change in Cushing Quality of Life (QoL) Normalized Total Score During the RW Phase
Description: The Cushing QoL patient questionnaire, which evaluates the health-related QoL in patients with Cushing syndrome, comprises 12 questions, each with 5 possible answers. The total score ranges from 12-60, with a higher score indicating improvement in QoL. The Cushing QoL instrument addresses known problem areas associated with Cushing syndrome including trouble sleeping, wound healing/bruising, irritability/mood swings/anger, self-confidence, physical changes, ability to participate in activities, interactions with friends and family, memory issues, and future health concerns.
Time Frame: Week 22 (end of OL Phase) and Week 36 (Week 12 of RW Phase)
Population: The analysis population was patients in the ITT-RW Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Relacorilant (RW Phase) | Placebo (RW Phase)
Number analyzed (Participants) | 27 | 31
score on a scale | 0.59 [-4.28 to 5.46] | -0.58 [-5.14 to 3.98]

10. Other Pre Specified Outcome: Percent Change in Tissue Fat Mass During the RW Phase
Description: Tissue fat mass was measured by dual energy X-ray absorptiometry (DXA) scan. Reported are change in in absolute tissue fat mass and change in percent tissue fat mass.
Time Frame: Week 22 (end of OL Phase) and Week 36 (Week 12 of RW Phase)
Population: The analysis population was patients in the ITT-RW Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Relacorilant (RW Phase) | Placebo (RW Phase)
Number analyzed (Participants) | 17 | 22
Percent Change
  Absolute Tissue Fat Mass | -0.64 [-1.684 to 0.400] | 1.67 [0.776 to 2.573]
  Percent Tissue Fat Mass | -0.14 [-1.031 to 0.759] | 1.66 [0.887 to 2.437]

11. Other Pre Specified Outcome: Number of Patients Who Worsened, as Assessed by the Global Clinical Response, During the RW Phase
Description: The Global Clinical Response assessment measures the patient's signs and symptoms of endogenous hypercortisolism in 7 clinical categories: 1) glucose parameters, 2) blood pressure parameters, 3) body composition parameters, 4) clinical appearance, 5) strength parameters, 6) psychiatric health/cognitive function parameters, and 7) quality of life using the Cushing QoL score. The overall response based on the totality of signs and symptoms is rated as +1 for improved, 0 for unchanged, and -1 for worsened. Each patient's final score is the median of ratings given by 3 members of the Data Review Board.
Time Frame: Week 22 (end of OL Phase) and up to Week 36 (Week 12 of RW Phase)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Percent Tissue Fat Mass During the OL Phase
Description: Tissue fat mass was measured by DXA scan.
Time Frame: Baseline and Week 22 (end of OL Phase)
Population: The analysis population was patients in the modified ITT-OL (mITT-OL) Population including all enrolled patients who received at least 1 dose of study drug and had at least 1 postbaseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Relacorilant (OL Phase)
Number analyzed (Participants) | 151
Percentage
  Baseline Percent Tissue Fat Mass: number analyzed (Participants) | 131
  Baseline Percent Tissue Fat Mass | 46.4 (8.39)
  Change from Baseline in Percent Tissue Fat Mass at Week 22: number analyzed (Participants) | 71
  Change from Baseline in Percent Tissue Fat Mass at Week 22 | -1.8 (2.73)

13. Other Pre Specified Outcome: Change in Cushing QoL Normalized Total Score During the OL Phase
Description: as for outcome 9
Time Frame: Baseline and Week 22 (end of OL Phase)
Population: The analysis population was patients in the mITT-OL Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relacorilant (OL Phase)
Number analyzed (Participants) | 151
score on a scale
  Baseline Cushing QoL Score | 41.9 (19.78)
  Change from Baseline in Cushing QoL Score: number analyzed (Participants) | 99
  Change from Baseline in Cushing QoL Score | 7.4 (14.63)

14. Other Pre Specified Outcome: Change in Beck Depression Inventory-II (BDI-II) Score During the OL Phase
Description: The BDI-II is a 21-question self-report inventory that measures depression. Each answer is scored with values of 0 to 3. The total score ranges from 0 to 63. Scores of 0 to 13 indicate minimal depression, 14 to 19; mild depression; 20 to 28; moderate depression; 29 to 63; severe depression.
Time Frame: Baseline and Week 22 (end of OL Phase)
Population: The analysis population was patients in the mITT-OL Population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Relacorilant (OL Phase)
Number analyzed (Participants) | 151
score on a scale
  Baseline BDI-II Score | 16.0 (10.24)
  Change from Baseline in BDI-II Score at Week 22: number analyzed (Participants) | 99
  Change from Baseline in BDI-II Score at Week 22 | -2.8 (8.91)

15. Other Pre Specified Outcome: Mean Change From Baseline in Body Weight During the OL Phase
Time Frame: Baseline and Week 22 (end of OL Phase)
Population: The analysis population was patients in the mITT-OL Population.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Relacorilant (OL Phase)
Number analyzed (Participants) | 151
kg
  Baseline Body Weight | 93.82 (24.734)
  Change from Baseline in Body Weight at Week 22: number analyzed (Participants) | 97
  Change from Baseline in Body Weight at Week 22 | -3.31 (5.861)

16. Other Pre Specified Outcome: Change in 2-hour Plasma Glucose During the OL Phase
Description: Plasma glucose was measured using the 2-hour oGTT.
Time Frame: Baseline and Week 22 (end of OL Phase)
Population: The analysis population was patients in the mITT-OL Population who had DM/IGT with or without HTN at Baseline.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Relacorilant (OL Phase)
Number analyzed (Participants) | 120
mmol/L
  Baseline oGTT: number analyzed (Participants) | 119
  Baseline oGTT | 14.370 (4.9402)
  Change from Baseline in oGTT at Week 22: number analyzed (Participants) | 71
  Change from Baseline in oGTT at Week 22 | -2.117 (4.6354)

17. Other Pre Specified Outcome: Change in Hemoglobin HbA1c During the OL Phase
Time Frame: Baseline and Week 22 (end of OL Phase)
Population: The analysis population was patients in the mITT-OL Population who had DM/IGT at Baseline.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Relacorilant (OL Phase)
Number analyzed (Participants) | 120
Percentage
  Baseline HbA1c | 7.16 (1.626)
  Change from Baseline in HbA1c at Week 22: number analyzed (Participants) | 74
  Change from Baseline in HbA1c at Week 22 | -0.29 (1.014)

18. Other Pre Specified Outcome: Change in SBP and DBP During the OL Phase
Description: Blood pressure was measured by 24-hour ABPM.
Time Frame: Baseline and Week 22 (end of OL Phase)
Population: The analysis population was patients in the mITT-OL Population who had HTN at Baseline.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Relacorilant (OL Phase)
Number analyzed (Participants) | 102
mm Hg
  Baseline SBP: number analyzed (Participants) | 101
  Baseline SBP | 140.66 (10.66)
  Change from Baseline in SBP at Week 22: number analyzed (Participants) | 66
  Change from Baseline in SBP at Week 22 | -7.9 (9.78)
  Baseline DBP: number analyzed (Participants) | 101
  Baseline DBP | 88.9 (7.20)
  Change from Baseline in DBP at Week 22: number analyzed (Participants) | 66
  Change from Baseline in DBP at Week 22 | -5.4 (6.98)

ADVERSE EVENTS:
Time Frame: OL Phase: Up to 22 weeks; RW Phase: up to 18 weeks after completion of the OL Phase.
Arm/Group | Relacorilant (OL Phase) | Relacorilant (RW Phase) | Placebo (RW Phase)
All-Cause Mortality (participants affected / at risk) | 2/152 | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 29/152 | 5/30 | 1/32
Other Adverse Events (participants affected / at risk) | 147/152 | 22/30 | 27/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relacorilant (OL Phase) (N=152) | Relacorilant (RW Phase) (N=30) | Placebo (RW Phase) (N=32)
Bone abscess (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0
Cavernous sinus thrombosis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Epididyitis (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Sinusitis fungal (Infections and infestations) | 1 | 0 | 0
Staphylococcal osteomyelitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Wound abscess (Infections and infestations) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Eye oedema (Eye disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Granuloma (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Congenital mitral valve incompetence (Congenital, familial and genetic disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relacorilant (OL Phase) (N=152) | Relacorilant (RW Phase) (N=30) | Placebo (RW Phase) (N=32)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 41 | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 17 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 52 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 28 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 23 | 0 | 0
Constipation (Gastrointestinal disorders) | 23 | 0 | 0
Vomiting (Gastrointestinal disorders) | 19 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 17 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 8 | 0 | 0
Oedema peripheral (General disorders) | 50 | 2 | 1
Fatigue (General disorders) | 34 | 0 | 0
Asthenia (General disorders) | 19 | 0 | 0
Peripheral swelling (General disorders) | 15 | 0 | 0
Pain (General disorders) | 13 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 31 | 3 | 4
Dizziness (Nervous system disorders) | 23 | 0 | 0
Paraesthesia (Nervous system disorders) | 21 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 13 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 24 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 12 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 0 | 0
Urinary tract infection (Infections and infestations) | 11 | 0 | 0
COVID-19 (Infections and infestations) | 9 | 2 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 17 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 0 | 0
Hypotension (Vascular disorders) | 10 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 12 | 0 | 4
Irritability (Psychiatric disorders) | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 1 | 2
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 2 | 0
Blood pressure increased (Investigations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual publications will be allowed before publication of the multicenter results, except as agreed with the Sponsor. The Investigator agrees to submit all manuscripts or abstracts to the Sponsor for review before submission to the publisher.

DOCUMENTS (2):
  • Study Protocol (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT03697109/Prot_002.pdf
  • Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT03697109/SAP_001.pdf